CLINICAL TRIAL: NCT03445416
Title: Increasing Healthcare Engagement Via Routine Vaccination Among Young Black Men Who Have Sex With Men
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not funded and therefore never began.
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Northwestern University (Other); Florida State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PA18162
Record Dates: First submitted 2018-02-03; First posted 2018-02-26 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Meningitis; HPV - Anogenital Human Papilloma Virus Infection; Hepatitis A
MeSH Terms: conditions — Meningitis; Hepatitis A

STUDY DESIGN:
Intervention Model Description: We will employ an experimental design with pre/posttest measures to determine changes in vaccination awareness, intention and status, as well as engagement in health care. A total of 20 POLs will be identified and randomized to either the intervention or comparison arm. Regardless of assignment, POLs will be asked to diffuse information to at least 5 YBMSM network recruits; either the intervention (comprised of vaccination messaging developed in partnership with YBMSM) or comparison group health messaging. The comparison group content will be developed by the investigative team and consist of general, non-tailored health-related messaging (e.g., no vaccination messaging, will not address stigma or medical mistrust). Outcome analysis will compare the 50 intervention recruits to the 50 SOC recruits at 3 months post intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: POL arm (Experimental): POL intervention. Enrolled POLs will be randomized at their intake visit; those randomized to the intervention arm will attend the popular opinion leader training (developed in Aim 1) and will be asked to diffuse the intervention messages to their network recruits.
  Interventions: Behavioral: POL arm
- Comparison group (Active Comparator): POLs who are randomized to the comparison arm will receive an abbreviated version of the POL training that includes general health messaging, but does not incorporate medical mistrust, stigma or specific vaccination messaging.
  Interventions: Behavioral: Comparison arm

INTERVENTIONS:
Behavioral: POL arm — A popular opinion leader intervention designed to increase routine vaccination among young black men who have sex with men.
  Arms: Intervention: POL arm
Behavioral: Comparison arm — A popular opinion leader intervention designed to increase routine vaccination among young black men who have sex with men.
  Arms: Comparison group

SUMMARY:
Vaccine-preventable diseases such as hepatitis A and meningitis, as well as cancers caused by human papillomavirus (HPV) disproportionately impact young Black men who have sex with men (YBMSM). Traditional techniques of vaccination promotion have been unable to address the racial disparities in vaccination rates. One promising method for influencing behavior change within YBMSM networks is diffusion of information through Popular Opinion Leaders (POLs). The POL model engages persons who are leaders within their own networks/communities to promote behavior change. The objective of this project is to develop and pilot test a POL intervention to increase routine HAV, HPV and meningococcal conjugate vaccination among YBMSM, ages 18-26. research (PAR) framework to facilitate community support and ensure intervention strategies are salient. PAR includes community members as equal collaborators in the research process. Outcomes from these aims are expected to have an impact on health outcomes by identifying effective strategies for increasing vaccination and routine healthcare engagement among YBMSM.

DETAILED DESCRIPTION:
For young black men who have sex with men (YBMSM), being at the intersection of racial and sexual minority status negatively impacts their access to healthcare and health seeking behavior, both of which fuel health disparities-particularly in infectious diseases. Prominent illustrations of these health disparities can be seen in reduced healthcare engagement and receipt of recommended vaccinations. Vaccine-preventable diseases such as hepatitis A and meningitis, as well as cancers caused by human papillomavirus (HPV) disproportionately impact MSM. As such, MSM are considered to be at high risk and are recommended to receive routine vaccination for hepatitis A (HAV), human papillomavirus (HPV) and meningitis. However, very little is known about how to promote uptake of routine vaccination among YBMSM. Traditional techniques of vaccination promotion (e.g., leveraging healthcare providers, school entry requirements) have been unable to address the racial disparities in vaccination rates. One promising method for influencing behavior change within YBMSM networks is diffusion of information through Popular Opinion Leaders (POLs). Trusted POLs may be successful in mitigating barriers in which traditional approaches have failed. The POL model engages persons who are leaders within their own networks/communities to promote behavior change. In response to PA-18-162 ("Health Promotion among Racial and Ethnic Minority Males"), the objective of this project is to develop and pilot test a POL intervention to increase routine HAV, HPV and meningococcal conjugate vaccination among YBMSM, ages 18-26. The long-term goal of our research is to reduce health disparities by identifying effective strategies to engage YBMSM in preventive healthcare. YBMSM will be included in all phases of research via a participatory action research (PAR) framework to facilitate community support and ensure intervention strategies are salient. PAR includes community members as equal collaborators in the research process. Outcomes from these aims are expected to have an impact on health outcomes by identifying effective strategies for increasing vaccination and routine healthcare engagement among YBMSM.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* report a social or sexual connection to at least 15 YBMSM
* be willing to diffuse information through their networks
* score at least 25 on the opinion leadership scale
* live in the Chicago area
* be available for the POL training

Exclusion criteria:

* Younger than age 18
* Less than 15 YBMSM in network
* Score lower than 25 on leadership scale
* Live outside the Chicago area
* Not available for the POL training

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Must identify as male
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Change in vaccine awareness | baseline, 3 months
  Participant reports increased awareness of preventative vaccines

SECONDARY OUTCOMES:
Change in vaccine status abstracted from medical record | baseline, 3 months
  HPV, meningococcal conjugate and HAV vaccination status of participant
Change in healthcare engagement | baseline, 3 months
  Number of doctor visits; access to primary care

CONTACTS AND LOCATIONS:
Overall Officials: Amy K Johnson, PhD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago

IPD SHARING:
Plan to Share IPD: No